CLINICAL TRIAL: NCT04593849
Title: Therapeutic Effects of Topical Herbal Medicine on Upper Extremities Fracture
Brief Title: Therapeutic Effects of Traditional Chinese Medicine in Topical Use on Upper Extremities Fracture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: YUAN-CHIEH YEH (Other)
Responsible Party: Sponsor-Investigator, YUAN-CHIEH YEH, Deputy director of traditional chinese medicine department, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202001174A3
Record Dates: First submitted 2020-10-09; First posted 2020-10-20 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Bone Fractures; Traditional Chinese Medicine; Chinese Herbal Medicine
Keywords: Wan Yin Gao; Chinese herbal patch; Upper Extremity fracture; Ru Yih Jin Huang Saan; Chinese herbal ointment; Wan Yin Gao Jia Jean Wey; Upper Extremities Fracture; Traditional Chinese Medicine; Chinese herbal medicine
MeSH Terms: conditions — Fractures, Bone | interventions — Pharmaceutical Preparations; Therapeutic Uses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Ru-Yih-Jin- Huang-Saan group) (Active Comparator): Herbal medicine(Ru-Yih-Jin- Huang-Saan) will be applied to injured site and covered with gauze for 6 hours per day. Each subject will receive persistent treatment for 1 week
  Interventions: Other: Ru-Yih-Jin- Huang-Saan(RYJHS), Wan-Yin-Gao-Jia-Jean-Wey(WYGJJW), placebo ( topical agent without therapeutic effects)
- group B (Wan-Yin-Gao-Jia-Jean-Wey group) (Experimental): Herbal medicine (Wan-Yin-Gao-Jia-Jean-Wey) will be applied to injured site and covered with gauze for 6 hours per day. Each subject will receive persistent treatment for 1 week
  Interventions: Other: Ru-Yih-Jin- Huang-Saan(RYJHS), Wan-Yin-Gao-Jia-Jean-Wey(WYGJJW), placebo ( topical agent without therapeutic effects)
- placebo group( topical agent without therapeutic effects) (Placebo Comparator): topical agent without therapeutic effects will be applied to injured site and covered with gauze for 6 hours per day. Each subject will receive persistent treatment for 1 week
  Interventions: Other: Ru-Yih-Jin- Huang-Saan(RYJHS), Wan-Yin-Gao-Jia-Jean-Wey(WYGJJW), placebo ( topical agent without therapeutic effects)
- control group (No Intervention): only oral analgesics will be applied to patients

INTERVENTIONS:
Other: Ru-Yih-Jin- Huang-Saan(RYJHS), Wan-Yin-Gao-Jia-Jean-Wey(WYGJJW), placebo ( topical agent without therapeutic effects) — We conduct a clinical trial using topical herbal medicine, including Ru-Yih-Jin- Huang-Saan(RYJHS) and Wan-Yin-Gao-Jia-Jean-Wey (WYGJJW) in treating post fracture pain and tissue swell. 24 eligible participants diagnosed of upper limb fracture with soft tissue injury grading of C1, C0 from Tscherne classification transferred from Orthopedic outpatient clinic and inpatient will be enrolled and randomly allocated to 4 groups, including experimental group A (RYJHS group), group B (WYGJJW group), placebo group( topical agent without therapeutic effects), and control group (only oral analgesics group), with 6 participants in each group.
  Arms: group A (Ru-Yih-Jin- Huang-Saan group); group B (Wan-Yin-Gao-Jia-Jean-Wey group); placebo group( topical agent without therapeutic effects)

SUMMARY:
There is no study evaluating the clinical effect of traditional chinese medicine(TCM) in topical use on musculotendinous injury, nor is that investigating the effectiveness on bone fracture healing. We hypothesize that with aid of topical chinese herbal medicine in addition to oral analgesics can be more beneficial in treating post traumatic injury, launching early mobilization, and enhancing fracture healing process.

DETAILED DESCRIPTION:
Orthopedic fractures are a common acute health issue, which often accompanied with life-long burden, accounts up to 34% total lifetime medical costs in the United States. It may also lead to significant long-term morbidity and, potentially, mortality if treated Improperly. Initial management is particularly crucial in helping the bone fracture healing process and reducing comorbidity. Apart from fracture fixation through nonoperative/conservative or operative methods in aim to restore anatomic alignment, oral analgesics are same important in Orthopedics patients in symptomatic control and for early mobilization. Non-opioid medication such as Acetaminophen or NSAIDs are routinely used for injury or postoperative pain management, despite that inevitable side effects including gastrointestinal bleeding and inconsistent show concerns of NSAIDs impairing bone healing in historical animal-based studies.

In which case, topical agents used in traditional chinese medicine(TCM) usually become a well-placed supplement to relieve inflammatory conditions. In spite of the lack of scientific evidence of efficacy, topical applications such as Ru- Yih-Jin-Huang-Saan (RYJHS) and Wan-Yin-Gao(WYG) have been used on musculoskeletal injuries in oriented countries for centuries, as their transcutaneous transport of the herbal chemicals to deeper tissues show biological activities of anti-inflammation, reducing swelling soft tissue, angiogenesis, fracture healing and cellular proliferation.

To date, there is no study evaluating the clinical effect of traditional chinese medicine in topical use on musculotendinous injury, nor is that investigating the effectiveness on bone fracture healing. We hypothesize that with aid of topical chinese herbal medicine in addition to oral analgesics can be more beneficial in treating post traumatic injury, launching early mobilization, and enhancing fracture healing process.

ELIGIBILITY:
Inclusion Criteria:

* Aged above 18 years with upper extremity fractures, including clavicle fractures, humerus fractures, forearm fractures, carpal bone fractures, finger fractures, etc.
* simple fractures with non-displacement or mild displacement, including transverse fracture, oblique fracture, linear fracture, impacted fracture, etc
* no need for surgery according to the orthopedist's evaluation
* willing to sign the informed consent of study and can cooperate with the doctor
* According to the orthopedist's evaluation, the soft tissue injury was grade C0 or C1 by Tscherne classification and without a high risk of infection

Exclusion Criteria:

* Compound fractures
* Simple fractures with moderate displacement or severe displacement
* The fracture pattern was a simple fracture but unstable, such as communicated fracture, etc.
* need for surgery according to the orthopedist's evaluation
* there were open wounds or at a high risk of infection
* According to the orthopedist's evaluation, the soft tissue was grade C2 or above by Tscherne classification and at a high risk of infection
* Unable to complete the questionnaire or cooperate with the doctor
* Allergy to Chinese herbal medicine patch or ointment
* Pregnancy
* heavy smoker
* Systemic diseases such as severe anemia, thyroid disease, uncontrolled diabetes mellitus, etc.
* Patients already on other treatment for upper extremity fractures, such as acupuncture therapy or transcutaneous electrical nerve stimulation
* Using other Chinese herbal medicine patch or ointment for treating upper extremity fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
reduction of pain | 1 week
  quantified by Visual Analogue Scale scoring system, Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain", providing a range of scores from 0-100 [100-mm scale]. A higher score indicates greater pain intensity.
swelling | 1 week
  recording circumference at the swelling site by tape measure
absence of adverse skin reaction to topical medicine | 1 week
  scored with Dyshidrotic Eczema Area and Severity Index (DASI index). The total score of the DASI results from the sum of severity grade score points of each of the four items (V = vesicles, E = erythema, S = desquamation, I = itch) multiplied by the affected area (A) score points: DASI = (pV + pE + pS + pI) × pA.
  The maximum possible score is 60. By the DASI, the dyshidrotic eczema is graded as: mild (0-15), moderate (16-30) and severe (31-60).

SECONDARY OUTCOMES:
improvement of functional performances | 1 week
  calculated by The Disabilities of the Arm, Shoulder and Hand Score (QuickDash), ranging from 0 (no disability) to 100 (most severe disability)
recovery of bone alignment and union at the fracture site | 1 week
  validated with radiographic images

CONTACTS AND LOCATIONS:
Locations (1):
- Keelung Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Derived] Lin WY, Lu CA, Chang CW, Yeh YC. Therapeutic Effects of Topical Traditional Chinese Medicine on Upper Extremity Fractures. Int J Gen Med. 2025 Jun 9;18:2973-2988. doi: 10.2147/IJGM.S511294. eCollection 2025. PMID 40520457